CLINICAL TRIAL: NCT04842188
Title: Evaluation of Leukocyte Platelet Rich Fibrin With Antimicrobial Photodynamic Therapy in Treatment of Furcation Involvement: Randomised Clinical Study
Brief Title: Furcation Treatment With L-PRF and aPDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, lecturer of oral medicine and periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: elamrousy2020
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Furcation Defects
Keywords: platelet rich fibrin; photodynamic therapy
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF (Active Comparator): Leukocyte platelet rich fibrin as a sole graft material in class II furcation
  Interventions: Procedure: L-PRF
- L-PRF with aPDT (Active Comparator): Leukocyte platelet rich fibrin combined with antibacterial photodynamic therapy in class II furcation
  Interventions: Procedure: L-PRF with aPDT

INTERVENTIONS:
Procedure: L-PRF with aPDT — surgical open flap debridement followed by L-PRF with aPDT
  Arms: L-PRF with aPDT
Procedure: L-PRF — surgical open flap debridement followed by L-PRF alone
  Arms: L-PRF

SUMMARY:
To treat grade II periodontally diseased furcation areas Leukocyte-Platelet Rich Fibrin (L-PRF) combined with antimicrobial Photo-Dynamic Therapy (a-PDT) was used.

DETAILED DESCRIPTION:
randomized, triple-blinded study (patient, clinician and biostatistician). Twenty-four patients with Grade II furcation involvement were recruited in this study.

Control group only received L-PRF, while study group used a combination of L-PRF and aPDT Attachment level, pocket depth, horizontal component and gingival recession, also radiographic Bone depth, width, height and volume were were recorded at baseline and postoperatively after 6 months

ELIGIBILITY:
Inclusion Criteria:

* Grade II furcation involvement
* age range 18- 50 years
* 3 mm or more vertical probing depth

Exclusion Criteria:

* systemic disease
* abnormal clotting and bleeding
* smokers,
* root caries or restoration
* Grade II mobility
* periapical lesions

Ages: 32 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of Vertical clinical attachment level VCAL | 6 months
  using periodontal probe in mm
clinical evaluation of vertical pocket depth VPD | 6 months
  using periodontal probe in mm
clinical evaluation of furcation horizontal component FHC | 6 months
  using periodontal probe in mm
clinical evaluation of gingival recession REC | 6 months
  using periodontal probe in mm

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No